CLINICAL TRIAL: NCT01371786
Title: A Phase 1, Open Label, Two Period, Randomized, Cross Over Scintigraphy Study Assessing Nasal Deposition of a Single Dose of a Ciclesonide Radiolabeled Solution Following Nasal Inhalation of a Novel Nasal Metered Dose Inhaler (MDI) and of a Mometasone Furoate Monohydrate Radiolabeled Suspension Via an Aqueous (AQ) Nasal Spray
Brief Title: A Phase 1 Scintigraphy Study to Assess Nasal Deposition of Ciclesonide. Using a Novel Nasal Metered Dose Inhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060-102
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Rhinitis (AR)
Keywords: Ciclesonide; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ciclesonide nasal aerosol (Experimental): A radiolabeled solution of ciclesonide nasal aerosol supplied in a 37 μg/actuation canister followed by a washout period of 120 hours and a radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle
  Interventions: Drug: ciclesonide nasal aerosol
- mometasone (Active Comparator): A radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle followed by a washout period of 120 hours and a radiolabeled solution of ciclesonide nasal aerosol supplied in a 37 μg/actuation canister
  Interventions: Drug: mometasone Aqueous (AQ) nasal spray

INTERVENTIONS:
Drug: ciclesonide nasal aerosol — A radiolabeled solution of ciclesonide nasal aerosol supplied in a 37 μg/actuation canister
  Arms: ciclesonide nasal aerosol
Drug: mometasone Aqueous (AQ) nasal spray — A radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle
  Arms: mometasone

SUMMARY:
This study is an open label, single dose, single site, randomized, cross over study that will assess nasal deposition of radioactivity following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal Metered Dose Inhaler (MDI) and of a mometasone furoate monohydrate radiolabeled suspension via an aqueous nasal spray in approximately 10-14 patients with symptomatic allergic rhinitis, aged 18-65 years.

DETAILED DESCRIPTION:
This study is an open label, single dose, single site, randomized, cross over study that will assess nasal deposition of radioactivity following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and of a mometasone furoate monohydrate radiolabeled suspension via an aqueous nasal spray in approximately 10 14 patients with symptomatic allergic rhinitis, aged 18 65 years. In order to ensure that patients will be symptomatic at the time of dosing, participants will be asked to withhold their usual treatments for perennial or seasonal allergic rhinitis, beginning at the Screening Visit until after Study Visit 3.

Each patient will be randomly assigned to one of two treatment sequences. The two treatments in this study are a single dose (one 37 mcg actuation per nostril) of radiolabeled solution of ciclesonide nasal aerosol 74 µg (Regimen A) and a single dose (two 50 mcg actuations per nostril) of a radiolabeled suspension of mometasone aqueous nasal spray 200 µg (Regimen B).

ELIGIBILITY:
Inclusion Criteria:

* Patient has give written informed consent and agrees to adhere to concomitant medication withholding periods, prior to participation.
* Patient is aged 18-65 years, inclusive.
* Patient has a Body Mass Index (BMI) of 18-30 kg/m2, inclusive
* Patient must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, medical history, and clinical laboratory values (Hematology, Chemistries and Urinalysis).
* A history of perennial or seasonal allergic rhinitis confirmed on GP report, or clinical diagnosis of perennial or seasonal allergic rhinitis confirmed at screening.
* A demonstrated sensitivity at the Screening visit, or within the 90 days prior to screening, to at least one allergen known to induce PAR (house dust mite, animal dander, cockroach, and molds) or SAR (grass pollen, tree pollen and weed pollen) using a 3 mm response to a standard skin prick test. The patient's positive allergen test must be consistent with the medical history of PAR/SAR.
* Must be willing and able to communicate and participate in the whole study.
* Patients must refrain from taking medication for allergic rhinitis, from Screening until completion of second dosing period.
* Patients, if female, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

  1. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation.
  2. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  3. True abstinence, when this is in line with the preferred and usual lifestyle of the patient (if the patient is usually not sexually active but becomes active, they with their partner, must use an acceptable method of birth control).

Exclusion Criteria:

* Female patient who is pregnant or lactating.
* Patient has radiation exposure from clinical trials, including that from the present study, excluding background radiation but including diagnostic X rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
* Patient has an abnormality on physical examination that, in the investigator's opinion, would affect nasal airway resistance, including: nasal jewelry or piercings; nasal pathology such as nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; or nasal ulcers or perforations.
* Patient has a history of cocaine or glue sniffing.
* Nasal surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the last 60 days prior to the Screening visit.
* Patient is a smoker (based on results of breath carbon monoxide testing at screening; ie, ≥10 ppm).
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta agonists and any controller drugs (eg, theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta agonists is acceptable. Use of short acting beta agonists for exercise induced bronchospasm will be allowed.
* Patient has a history of any chronic respiratory disorder including active or quiescent pulmonary tuberculosis.
* Patient has a history of adverse reaction or allergy to ciclesonide, mometasone, other corticosteroids, or formulation excipients.
* Patient has a Screening forced expiratory volume (FEV1) <80% of the predicted value for their age, sex, height and race.
* Patient has had an upper respiratory tract infection (excluding otitis media) within 14 days of first dosing period, or a lower respiratory tract infection within 3 months of the first study day.
* Previous participation in an intranasal ciclesonide HFA nasal aerosol study; participation in any investigational drug trial within the 60 days preceding the Screening visit or planned participation in another investigational drug trial at any time during this trial.
* History of alcohol or drug abuse within 2 years preceding the Screening visit.
* Study participation by clinical investigator site employees and/or their relatives or by more than one patient from the same household.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the patients availability to participate in the clinical trial:

  * impaired hepatic function including alcohol related liver disease or cirrhosis
  * history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts
  * any systemic infection including a history of a positive test for HIV, hepatitis B or hepatitis C.
  * hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism)
  * gastrointestinal disease
  * malignancy (excluding basal cell carcinoma)
  * current neuropsychological condition with or without drug therapy
  * Any condition that, in the judgment of the investigator, would preclude the patient from completing the protocol with capture of the assessments as written.
  * Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington Fields, Ruddington, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence Ciclesonide Nasal Aerosol /Mometsasone Aqueous: A radiolabeled solution of ciclesonide nasal aerosol supplied in a 37 μg/actuation canister followed by a washout period of 120 hours and a radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle
- Sequence Mometasone Aqueous / Ciclesonide Nasal Aerosol: A radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle followed by a washout period of 120 hours and a radiolabeled solution of ciclesonide nasal aerosol supplied in a 37 μg/actuation canistermometasone Aqueous (AQ) nasal spray : A radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle
- Total: Total of all reporting groups
Arm/Group | Sequence Ciclesonide Nasal Aerosol /Mometsasone Aqueous | Sequence Mometasone Aqueous / Ciclesonide Nasal Aerosol | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.1 (13.62) | 34.6 (11.96) | 35.4 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Initial Deposition of Radioactivity Within the Nasal Cavity as a Percent of Delivered Dose
Description: The scintigraphic measure of radioactivity initially deposited (approximately 2 minutes post-dose) within the nasal cavity, expressed as a percent of the delivered dose (i.e., the total amount of radioactivity delivered), following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and a mometasone radiolabeled suspension via an aqueous nasal spray.
Time Frame: Day 1 at 2 minutes post dose
Population: Scintigraphic Population
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled
Groups:
- Mometasone: A radiolabeled suspension of mometasone Aqueous (AQ) nasal spray supplied in a 50 μg/actuation bottle
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Number analyzed (Participants) | 14 | 13
percentage of radiolabeled | 99.48 (0.98) | 86.28 (11.99)
Statistical Analysis 1: Comparison: Ciclesonide Nasal Aerosol vs Mometasone; No formal null hypothesis was stated or tested.Descriptive statistics only were calculated and presented. The sample size was determined outside of statistical considerations. The sample size of 10 subjects was sufficient to provide approximately 80% power to detect a difference of 25% between the two treatment groups in the percentage of nasal deposition approximately 2 minutes post dose, assuming a two-sided test evaluated at a significance level of 0.05, with a SD of the difference of 23.17%; Test type: Superiority or Other; No formal statistical testing was conducted. Only descriptive statistics were calculated and presented; Mean Difference (Final Values) = -12.92, 95% CI 2-sided [-21.76 to -4.09] — Difference calculated as Mometasone minus Ciclesonide

2. Secondary Outcome: Initial Deposition of Radioactivity Within the Nasopharynx as a Percent of Delivered Dose
Description: The scintigraphic measure of radioactivity initially deposited (approximately 2 minutes post-dose) within the nasopharynx, expressed as a percent of the delivered dose (i.e., the total amount of radioactivity delivered), following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and a mometasone radiolabeled suspension via an aqueous nasal spray.
Time Frame: Day 1 at 2 minutes post-dose
Population: Scintigraphic Population
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Number analyzed (Participants) | 14 | 13
percentage of radiolabeled | 0.03 (0.11) | 1.58 (1.94)

3. Secondary Outcome: Deposition of Radioactivity Within the Nasal Cavity Over 10 Minutes as a Percent of Delivered Dose
Description: The scintigraphic measure of radioactivity deposited within the nasal cavity, expressed as a percent of the delivered dose (i.e., the total amount of radioactivity delivered), over 10 minutes (at approximately 2 minute intervals post-dose) following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and a mometasone radiolabeled suspension via an aqueous nasal spray.
Time Frame: Average of 2, 4, 6, 8 and 10 minutes post dose
Population: Scinitgraphic Population
Measure: Mean (Standard Deviation); unit: percentage of of radiolabled
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Number analyzed (Participants) | 14 | 13
percentage of of radiolabled | 89.61 (11.80) | 69.15 (18.08)

4. Secondary Outcome: Initial Deposition of Radioactivity on Nasal Wipes as a Percent of Delivered Dose
Description: The scintigraphic measure of radioactivity initially deposited (approximately 2 minutes post-dose) on nasal wipes, expressed as a percent of the delivered dose (i.e., the total amount of radioactivity delivered), following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and a mometasone radiolabeled suspension via an aqueous nasal spray.
Time Frame: Day 1 at 2 minutes post-dose
Population: Scintigraphic Population
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Number analyzed (Participants) | 14 | 13
percentage of radiolabeled | 0.49 (0.98) | 12.15 (12.83)

5. Secondary Outcome: Deposition of Radioactivity Within on Nasal Wipes Over 10 Minutes as a Percent of Delivered Dose
Description: The scintigraphic measure of radioactivity deposited on nasal wipes, expressed as a percent of the delivered dose (i.e., the total amount of radioactivity delivered), over 10 minutes (at approximately 2 minute intervals post-dose) following nasal inhalation of a ciclesonide radiolabeled solution via a novel nasal MDI and a mometasone radiolabeled suspension via an aqueous nasal spray.
Time Frame: Average of 2, 4, 6, 8, and 10 minutes post dose
Population: Scinitigraphic Population
Measure: Mean (Standard Deviation); unit: percentage of radiolabeled
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Number analyzed (Participants) | 14 | 13
percentage of radiolabeled | 0.98 (1.71) | 13.15 (12.63)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Ciclesonide Nasal Aerosol | Mometasone
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide Nasal Aerosol (N=14) | Mometasone (N=14)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Both the formulations used in this study were radiolabeled and not the individual corticosteroid molecules. Therefore the distribution of the corticosteroid molecules over 10 minutes post-administration was not quantified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other